CLINICAL TRIAL: NCT00627328
Title: The Atrial High Rate Episodes (A-HIRATE) in Pacemaker Patients
Brief Title: The Atrial High Rate Episodes in Pacemaker Patients
Status: Completed | Type: Observational
Sponsor: Medtronic Cardiac Rhythm and Heart Failure (Industry)
Responsible Party: Diane Sahr, CRDM Clincial Research
Other Study IDs: 163
Record Dates: First submitted 2007-12-26; First posted 2008-03-03 (Estimated); Last update posted 2008-03-03 (Estimated); Status verified 2008-02

CONDITIONS: Arrhythmia; Atrial Fibrillation; Atrioventricular Block; Bradycardia; Sick Sinus Syndrome
Keywords: Physiologic Pacing; Dual Chamber Pacing; Atrioventricular Block; Bradycardia; Sick Sinus Syndrome
MeSH Terms: conditions — Arrhythmias, Cardiac; Atrial Fibrillation; Atrioventricular Block; Bradycardia; Sick Sinus Syndrome

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- 1: pacemaker patients with previously diagnosed AT.
- 2: pacemaker patients without previously diagnosed AT.

SUMMARY:
Prospective study assessing the incidence of atrial high rate episodes (AHRE) in pacemaker patients with and without previously diagnosed AT.

DETAILED DESCRIPTION:
The purpose of this study is to assess the incidence of fast heart rates that originate in the upper chamber of the heart (atrial tachyarrhythmias) in pacemaker patients that have not been previously diagnosed with this condition. The study will also look at how the diagnostic feature in the pacemaker that detects atrial tachyarrhythmias helps physicians with the medical management of patients' heart rhythm.

ELIGIBILITY:
Inclusion Criteria:

* Patients undergoing a Medtronic Kappa DR 700 or Medtronic Kappa 900 DR implant, for approved indications
* No previous history of pacemaker implantation
* Patients 50 years of age or older

Exclusion Criteria:

* Patients with a history of atrial tachyarrhythmias (primary arm of study)
* Patients with medical conditions that would limit study participation
* Patients inaccessible for follow-up at the study center
* Patients incapable of providing Informed Consent
* Patients with NYHA classification of IV
* Patients with a history of neurocardiogenic syncope, long QT syndrome, or Hypertrophic Obstructive Cardiomyopathy (HOCM)
* Patients taking Sotalol or Amiodorone
* Patients with a history of a prior ICD or pacemaker implantation.

Min Age: 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Prospective study with patients undergoing a Medtronic Kappa DR 700 or Medtronic Kappa 900 DR implant, for approved indications.
Sampling Method: Non-Probability Sample
Enrollment: 427 (Actual)
Dates: Start 2000-07; Study Completion 2004-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: M. V. Orlov, MD, Principal Investigator — Tufts University School of Medicine; J.K. Ghali, MD, Principal Investigator — Louisiana State University Health Sciences Center in New Orleans
Locations (42):
- United States (37):
  - Hot Springs, Arkansas
  - Little Rock, Arkansas
  - Fresno, California
  - Glendale, California
  - San Diego, California
  - Daytona Beach, Florida
  - Orlando, Florida
  - Hammond, Indiana
  - Hobart, Indiana
  - Munster, Indiana
  - Louisville, Kentucky
  - Marrero, Louisiana
  - Shreveport, Louisiana
  - Salisbury, Maryland
  - West Roxbury, Massachusetts
  - Saint Cloud, Minnesota
  - Livingston, New Jersey
  - Patterson, New Jersey
  - Flushing, New York
  - Rochester, New York
  - Syracuse, New York
  - The Bronx, New York
  - Charlotte, North Carolina
  - Gastonia, North Carolina
  - Greenville, North Carolina
  - Willimington, North Carolina
  - Oklahoma City, Oklahoma
  - Bethlehem, Pennsylvania
  - Mechanicsburg, Pennsylvania
  - Scranton, Pennsylvania
  - Wynnewood, Pennsylvania
  - Providence, Rhode Island
  - Chattanooga, Tennessee
  - Dallas, Texas
  - Falls Church, Virginia
  - Richmond, Virginia
  - Milwaukee, Wisconsin
- Australia (3):
  - Ashford
  - Ballarat
  - Bedford Park
- France (2):
  - Lille
  - Rouen

REFERENCES:
- [Background] Ghali JK, Orlov MV, Araghi-Niknam M, Sherfesee L, Hettrick DA. The influence of symptoms and device detected atrial tachyarrhythmias on medical management: insights from A-HIRATE. Pacing Clin Electrophysiol. 2007 Jul;30(7):850-7. doi: 10.1111/j.1540-8159.2007.00772.x. PMID 17584266
- [Result] Orlov MV, Ghali JK, Araghi-Niknam M, Sherfesee L, Sahr D, Hettrick DA; Atrial High Rate Trial Investigators. Asymptomatic atrial fibrillation in pacemaker recipients: incidence, progression, and determinants based on the atrial high rate trial. Pacing Clin Electrophysiol. 2007 Mar;30(3):404-11. doi: 10.1111/j.1540-8159.2007.00682.x. PMID 17367361